CLINICAL TRIAL: NCT05040204
Title: The Effects of Dietary Supplementation on Serum Protein Glycosylation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 949221; 1K24AR077313-01A1 (NIH)
Record Dates: First submitted 2021-09-01; First posted 2021-09-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: dietary supplement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Supplement 1 (Experimental): 6 subjects will consume 12 grams of dietary supplement 1 daily for 4 weeks
  Interventions: Dietary Supplement: Monosaccharide Powder
- Experimental Supplement 2 (Experimental): 6 subjects will consume 12 grams of dietary supplement 2 daily for 4 weeks
  Interventions: Dietary Supplement: Monosaccharide Powder
- Experimental Supplement 3 (Experimental): 20 subjects will consume 50 grams of dietary supplement 3 daily for 4 weeks
  Interventions: Dietary Supplement: Monosaccharide Powder
- Placebo Comparator 1 (Placebo Comparator): 6 subjects will consume 12 grams of placebo dietary supplement daily for 4 weeks
  Interventions: Dietary Supplement: Placebo Comparator
- Placebo Comparator 2 (Placebo Comparator): 6 subjects will consume 50 grams of placebo dietary supplement daily for 4 weeks
  Interventions: Dietary Supplement: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Monosaccharide Powder — Monosaccharide powder dissolved in water.
  Arms: Experimental Supplement 1; Experimental Supplement 2; Experimental Supplement 3
Dietary Supplement: Placebo Comparator — Placebo (glucose powder)
  Arms: Placebo Comparator 1; Placebo Comparator 2

SUMMARY:
Two randomized double-blind placebo-controlled clinical studies to assess the effects of dietary glycan monomer supplementation on the immune system, especially antibody glycosylation in healthy adults. Immune profiling and glycoproteomics will be performed on serum isolated at these same time points.

ELIGIBILITY:
Inclusion Criteria:

* Adult men/women (age 18-45) who are in general good health with Body Mass Index (BMI) range of 18.5-25

Exclusion Criteria:

* Adults younger than 18 or older than 45 years of age
* Women who are pregnant, actively nursing or have had a pregnancy within the last year
* Women who are peri-menopausal or post-menopausal
* Women with irregular menstrual cycles (more frequently than every 21 days or lasts longer than 8 days. Missed, early, or late periods are also considered signs of an irregular cycle)
* Women on hormonal contraception, including birth control, hormonal intrauterine device, or contraceptive implant
* Individuals with past medical history of an autoimmune condition or malignancy, excluding non-melanoma skin cancer
* Individuals with cardiovascular, pulmonary, reproductive, endocrine, metabolic, neurologic, gastrointestinal, hematologic, or infectious diseases of any type
* Individuals with diagnosis of galactosemia or congenital disorders of glycosylation
* Individuals with phenylketonuria
* Individuals currently taking prescription medications, or who have taken prescription medications within the last 3 months
* Individuals currently taking over-the-counter medications
* Individuals currently taking or who have taken supplements including herbal, protein or vitamin supplements in the last 3 months (e.g. whey protein, St. John's Wort, green tea supplements, biotin, creatine supplements), excluding multivitamins or essential vitamins
* Individuals with BMI less than 18.5 or greater than 25
* Individuals with prior history of severe food or drug allergic reactions
* Individuals with allergic reaction or adverse reaction to shellfish, N-acetylglucosamine, galactose, Spirulina/chlorella/algae supplements, or arabinose containing compounds/foods/supplements
* Individuals with first-degree relative with history of an autoimmune condition
* Individuals with social history of current use of tobacco, alcohol or other drugs
* Individuals with dietary restrictions (vegetarians are permitted to participate in the study) or atypical exercise patterns, or to whom any of the following dietary habits or characteristics apply (the following exclusion criteria are placed to minimize variability in diet/exercise patterns in our pilot study population):
* Actively dieting or trying to lose weight
* Vegan diet
* Consume equal to or greater than 2 cups of tea a day
* Consume equal to or greater than 4 cups of coffee a day
* Consume equal to or greater than 3 cups of fruit juice a day
* Practice intensive exercise patterns (marathon training, workouts >4 hours a day)
* Consume soda or energy drinks of any amount
* Consume fast food equal to or greater than 5 days per week
* Consume greater than one serving of alcohol per day

  * (1 serving of wine = 6 oz, 1 serving of beer = 12 oz, 1 serving of spirits = 1 oz)
* On a carbohydrate-restricted or "Paleo" diet, or calorie-restricted diet (less than 20-25% of maintenance calories)
* Adults unable to consent
* Prisoners

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Characterize Immunoglobulin fragment crystallization modifications | 4 Weeks
  Use mass spectrometry and RNA sequencing from subject blood samples to characterize site specific glycosylation on Immunoglobulin A, Immunoglobulin M, and Immunoglobulin G.

SECONDARY OUTCOMES:
Assess for potential adverse events | 2 months after first dose
  Monitor symptoms, severity, and duration of adverse events.
Quantification of enzymatic modifications measured in grams by spectrometry | 6 months
  The investigators will measure enzymatic changes on glycoproteins in the immune system by spectrometry, i.e., these changes will be measured in grams. Spectometry will allow the investigators to quantify these changes in small detail, and therefore give a better idea of how supplementation can change enzymatic process that then affect the structure, and mass, of glycoproteins.
Flow cytometry to determine the effect of dietary supplementation on the immune system | 6 months
  Perform flow cytometry on subject blood samples to determine the effect of dietary supplement on immune system. For example, the investigators will note changes to immune cell pro-inflammatory and anti-inflammatory cytokine clusters as translated proteins (measured as height and area of cytokine intensity).
Transcriptome analysis to determine the effect of dietary supplementation on the immune system | 6 months
  Perform transcriptome analysis on subject blood samples to determine the effect of dietary supplement on immune system. For example, the investigators will note changes to immune cell pro-inflammatory and anti-inflammatory cytokine clusters as RNA (measure on a logarithmic scale per number of reads) to determine the effects of supplementation on both gene transcription and translation.

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/the-effects-of-dietary-supplementation-on-serum-protein-glycosylation-347100/